CLINICAL TRIAL: NCT03093506
Title: Effects of Micro-dose and Low-dose Recombinant Human Erythropoietin on Mitochondrial Function and Cognitive Performance
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Soeren Lundgaard Larsen, Physician, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-1-2011-098
Record Dates: First submitted 2015-01-08; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Human Volunteers
Keywords: Erythropoietin; Randomized controlled trial; Human volunteers; Mitochondrial function; Cognitive performance
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-dose rhEpo (Active Comparator): RhEpo 60IU/kg/week
  Interventions: Drug: Low-dose rhEpo
- Micro-dose rhEpo (Active Comparator): RhEpo 20IU/kg/week
  Interventions: Drug: Micro-dose rhEpo
- Placebo Control (Placebo Comparator): Saline
  Interventions: Other: Placebo Control

INTERVENTIONS:
Drug: Low-dose rhEpo — 60IU/kg/week
  Other Names: Recombinant Human Erythropoitin
  Arms: Low-dose rhEpo
Drug: Micro-dose rhEpo — 20IU/kg/week
  Other Names: Recombinant Human Erythropoitin
  Arms: Micro-dose rhEpo
Other: Placebo Control — Saline
  Other Names: Saline
  Arms: Placebo Control

SUMMARY:
A recent study by Plenge et al. revealed that rhEpo treatment enhances skeletal muscle mitochondrial respiratory capacity in humans indicating a muscle ergogenic effect of rhEpo on aerobic metabolism. The main purpose of the present study is to determine if a shorter treatment period with micro-dose as well as low-dose rhEpo has similar effects on muscle mitochondrial function.

Higher doses of rhEpo is known to increase cognitive performance, but it is not clear if lower doses of rhEpo have similar effects. A second purpose of the present study is to determine if micro-dose as well as low-dose rhEpo increases cognitive performance.

DETAILED DESCRIPTION:
Twenty-five healthy young male volunteers are randomized to either a low-dose rhEpo (60 IU/kg/week), micro-dose rhEpo (20 IU/kg/week), or placebo control (saline) group. All subjects receive two subcutaneous injections per week for four weeks. Muscle biopsies are taken at the beginning and end of the study period. Mitochondrial function is measured in permeabilized fibres using high-resolution respirometry with the substrates malate (2mM), octanoyl carnitine (1.5mM), glutamate (10mM), succinate (10mM), under saturating [ADP] (5mM), and with the membrane uncoupler FCCP (1μM).

On the first day before administration of rhEpo and after the four weeks' treatment the subjects are undergoing two cognitive performance-tests, Raven Standard Progressive Matrices (Raven), and Number Finder (NUFI). Weekly semi-structured interviews are conducted by a blinded interviewer focusing on experienced change in cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Normal medical examination
* Weekly exercise for 0-5 hours

Exclusion Criteria:

* Smoking daily
* Earlier use of performance-enhancing drugs
* Elite athletes
* Presence of cardiovascular or metabolic disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen-flux (picomol/second) | Four weeks

SECONDARY OUTCOMES:
Sum of speed-score and accuracy-score in the RAVEN-test | Four weeks
Number of correctly found fields in the NUFI-test | Four weeks
Rating of the interviews on a scale from -3 to +3 according to experienced change in ability to concentrate | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soeren L. Larsen, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Copenhagen University Hospital Bispebjerg, Department of Anaesthesiology, Copenhagen, Kbh NV, Denmark

REFERENCES:
- [Background] Plenge U, Belhage B, Guadalupe-Grau A, Andersen PR, Lundby C, Dela F, Stride N, Pott FC, Helge JW, Boushel R. Erythropoietin treatment enhances muscle mitochondrial capacity in humans. Front Physiol. 2012 Mar 13;3:50. doi: 10.3389/fphys.2012.00050. eCollection 2012. PMID 22419911
- [Derived] Viuff SL, Plenge U, Belhage B, Boushel R, Koester T. Effects of low-dose recombinant human erythropoietin treatment on cognitive performance. Dan Med J. 2017 Sep;64(9):A5403. PMID 28874242